CLINICAL TRIAL: NCT04806451
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of Crinecerfont (NBI-74788) in Pediatric Subjects With Classic Congenital Adrenal Hyperplasia, Followed by Open-Label Treatment
Brief Title: Global Safety and Efficacy Registration Study of Crinecerfont in Pediatric Participants With Classic Congenital Adrenal Hyperplasia (CAHtalyst Pediatric Study)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NBI-74788-CAH2006; 2020-004381-19 (EudraCT Number); 2023-509170-33-00 (EU CTIS Number)
Record Dates: First submitted 2021-03-16; First posted 2021-03-19 (Actual); Results first posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Congenital Adrenal Hyperplasia
Keywords: classic congenital adrenal hyperplasia (CAH); 21-hydroxylase deficiency
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital; Congenital adrenal hyperplasia due to 21 hydroxylase deficiency | interventions — crinecerfont

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Crinecerfont (Experimental): Crinecerfont solution or capsule, administered orally, twice daily for 28 weeks during the placebo-controlled treatment period, followed by active treatment with crinecerfont for at least 24 weeks.
  Interventions: Drug: Crinecerfont
- Placebo (Placebo Comparator): Placebo solution or capsule, administered orally, twice daily for 28 weeks, followed by active treatment with crinecerfont for at least 24 weeks.
  Interventions: Drug: Crinecerfont; Drug: Placebo

INTERVENTIONS:
Drug: Crinecerfont — CRF type 1 receptor antagonist
  Other Names: NBI-74788; Crenessity
Drug: Placebo — Non-active dosage form
  Arms: Placebo

SUMMARY:
This is a Phase 3 study to evaluate the efficacy, safety, and tolerability of crinecerfont versus placebo administered for 28 weeks in approximately 81 pediatric participants with classic congenital adrenal hyperplasia (CAH) due to 21-hydroxylase deficiency. The study consists of a 28-week double blind, placebo-controlled period, followed by 24 weeks of open-label treatment with crinecerfont. Subsequently, participants may elect to participate in the open-label extension (OLE) period. The duration of participation in the study is approximately 14 months for the core study and will be a variable amount of time per participant for the OLE (estimated to be approximately 3 years).

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to adhere to the study procedures, including all requirements at the study center, and return for the follow-up visit.
* Have a medically confirmed diagnosis of classic CAH due to 21-hydroxylase deficiency.
* Be on a stable steroid regimen.
* Have elevated androgen levels.
* Participants of childbearing potential must be abstinent or agree to use appropriate birth control during the study.

Exclusion Criteria:

* Have a diagnosis of any of the other forms of classic CAH.
* Have a history of bilateral adrenalectomy, hypopituitarism, or other condition requiring chronic glucocorticoid therapy.
* Have a clinically significant unstable medical condition or chronic disease other than CAH.
* Have a history of cancer unless considered to be cured.
* Have a known history of clinically significant arrhythmia or abnormalities on electrocardiogram (ECG).
* Have a known hypersensitivity to any corticotropin-releasing hormone antagonist.
* Have received an investigational drug within 30 days before initial screening or plan to use an investigational drug (other than the study drug) during the study.
* Have current substance dependence or substance (drug) or alcohol abuse.
* Have had a significant blood loss or donated blood or blood products within 8 weeks prior to the study.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 103 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2027-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Lead, Study Director — Neurocrine Biosciences
Locations (44):
- United States (22):
  - Neurocrine Clinical Site, Birmingham, Alabama
  - Neurocrine Clinical Site, Los Angeles, California
  - Neurocrine Clinical Site, Orange, California
  - Neurocrine Clinical Site, San Diego, California
  - Neurocrine Clinical Site, San Francisco, California
  - Neurocrine Clinical Site, Aurora, Colorado
  - Neurocrine Clinical Site, Hartford, Connecticut
  - Neurocrine Clinical Site, Washington D.C., District of Columbia
  - Neurocrine Clinical Site, Atlanta, Georgia
  - Neurocrine Clinical Site, Indianapolis, Indiana
  - Neurocrine Clinical Site, Boston, Massachusetts
  - Neurocrine Clinical Site, Ann Arbor, Michigan
  - Neurocrine Clinical Site, Minneapolis, Minnesota
  - Neurocrine Clinical site, St Louis, Missouri
  - Neurocrine Clinical Site, New Hyde Park, New York
  - Neurocrine Clinical Site, New York, New York
  - Neurocrine Clinical Site, Oklahoma City, Oklahoma
  - Neurocrine Clinical Site, Tulsa, Oklahoma
  - Neurocrine Clinical Site, Philadelphia, Pennsylvania
  - Neurocrine Clinical Site, Pittsburgh, Pennsylvania
  - Neurocrine Clinical Site, Dallas, Texas
  - Neurocrine Clinical Site, Seattle, Washington
- Belgium (2):
  - Neurocrine Clinical Site, Brussels
  - Neurocrine Clinical Site, Ghent
- Canada (3):
  - Neurocrine Clinical Site, Edmonton, Alberta
  - Neurocrine Clinical Site, Vancouver, British Columbia
  - Neurocrine Clinical Site, Montreal, Quebec
- France (4):
  - Neurocrine Clinical Site, Angers
  - Neurocrine Clinical Site, Bordeau
  - Neurocrine Clinical Site, Le Kremlin-Bicêtre
  - Neurocrine Clinical Site, Paris
- Germany (3):
  - Neurocrine Clinical Site, Berlin
  - Neurocrine Clinical Site, Heidelberg
  - Neurocrine Clinical Site, Magdeburg
- Neurocrine Clinical Site, Athens, Greece
- Italy (4):
  - Neurocrine Clinical Site, Bologna
  - Neurocrine Clinical Site, Milan
  - Neurocrine Clinical Site, Napoli
  - Neurocrine Clinical Site, Roma
- Poland (2):
  - Neurocrine Clinical Site, Gdansk
  - Neurocrine Clinical Site, Rzeszów
- Spain (2):
  - Neurocrine Clinical Site, Barcelona
  - Neurocrine Clinical Site, Seville
- Neurocrine Clinical Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sarafoglou K, Kim MS, Lodish M, Felner EI, Martinerie L, Nokoff NJ, Clemente M, Fechner PY, Vogiatzi MG, Speiser PW, Auchus RJ, Rosales GBG, Roberts E, Jeha GS, Farber RH, Chan JL; CAHtalyst Pediatric Trial Investigators. Phase 3 Trial of Crinecerfont in Pediatric Congenital Adrenal Hyperplasia. N Engl J Med. 2024 Aug 8;391(6):493-503. doi: 10.1056/NEJMoa2404655. Epub 2024 Jun 2. PMID 38828945

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study includes a double-blind (DB) placebo-controlled treatment period, an open-label (OL) treatment period, and an open-label extension (OLE) period. The OL treatment period and OLE period of the study is ongoing. Only the primary analysis results (as of 09 August 2023 data cutoff date) have been reported. The final results will be reported after completion of the study.
Groups:
- Placebo: Participants received crinecerfont-matched placebo orally twice daily for 28 weeks during the DB placebo-controlled treatment period. After the 28-week DB placebo-controlled treatment period, there was a 24-week, OL treatment period, during which all participants received crinecerfont at doses based on their Week 28 body weight.
- Crinecerfont: Participants received crinecerfont orally twice daily for 28 weeks during the DB placebo-controlled treatment period. Dose assignment from Day 1 to Week 28 was based on the participant's weight at Day 1. After the 28-week DB placebo-controlled treatment period, there was a 24-week, OL treatment period, during which all participants received crinecerfont at doses based on their Week 28 body weight.
Period: DB Treatment Period (28 Weeks)
Arm/Group | Placebo | Crinecerfont
Started | 34 | 69
Received at Least 1 Dose of Study Drug | 33 | 69
Completed | 31 | 66
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Adverse Event | 0 | 2
Period: OL Treatment Period (24 Weeks)
Arm/Group | Placebo | Crinecerfont
Started | 31 | 66
Received at Least 1 Dose of Study Drug | 31 | 66
Completed | 15 | 29
Not Completed | 16 | 37
Not completed — Ongoing in the Study | 16 | 37

BASELINE CHARACTERISTICS:
Population: Full Analysis Set included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Crinecerfont | Total
Number analyzed (Participants) | 34 | 69 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.142 (3.690) | 12.022 (3.405) | 12.061 (3.484)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 34 | 50
  Male | 18 | 35 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 8 | 11
  Not Hispanic or Latino | 25 | 52 | 77
  Unknown or Not Reported | 6 | 9 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 1 | 1
  Race: Asian | 2 | 7 | 9
  Race: Black or African American | 0 | 3 | 3
  Race: White | 23 | 42 | 65
  Race: Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Race: Other | 2 | 3 | 5
  Race: Multiple | 1 | 3 | 4
  Race: Not Collected | 6 | 9 | 15
Serum Androstenedione Concentration [Mean (Standard Deviation); unit: nanograms (ng)/deciliter (dL)] | 483.32 (455.64) | 404.96 (464.10) | 430.83 (460.58)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Serum Androstenedione at Week 4
Description: Blood serum samples were collected for the analysis of serum androstenedione concentrations. Least square (LS) mean and standard error (SE) were calculated using analysis of covariance (ANCOVA) model.
Time Frame: Baseline, Week 4
Population: Full Analysis Set included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: ng/dL
Arm/Group | Placebo | Crinecerfont
Number analyzed (Participants) | 34 | 69
ng/dL | 70.986 (56.198) | -196.789 (39.369)
Statistical Analysis 1: Comparison: Placebo vs Crinecerfont; Test type: Superiority; p = 0.0002, ANCOVA; LS Mean Difference = -267.775, 95% CI 2-sided [-403.427 to -132.124], Standard Error of Mean 68.313

2. Secondary Outcome: Change From Baseline in Serum 17-hydroxyprogesterone (17-OHP) at Week 4
Time Frame: Baseline, Week 4
Reporting Status: Not Posted

3. Secondary Outcome: Percent Change From Baseline in Glucocorticoid Daily Dose at Week 28
Time Frame: Baseline, Week 28
Reporting Status: Not Posted

4. Secondary Outcome: Number of Participants Who Achieved a Reduction to Physiologic Glucocorticoid Dose While Maintaining Androstenedione Control at Week 28
Time Frame: Week 28
Reporting Status: Not Posted

5. Secondary Outcome: Change From Baseline in Body Mass Index (BMI) Standard Deviation Score (SDS) at Week 28
Time Frame: Baseline, Week 28
Reporting Status: Not Posted

6. Secondary Outcome: Change From Baseline in Mean 24-hour Salivary 17-OHP at Week 28
Time Frame: Baseline, Week 28
Reporting Status: Not Posted

7. Secondary Outcome: Change From Baseline in the Ratio of Bone Age to Chronological Age (BA:CA) at Week 28
Time Frame: Baseline, Week 28
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Baseline up to Week 28
Description: Per planned analysis all-cause mortality data were collected and reported for all randomized participants. Adverse events (serious and other) were collected and reported for all randomized participants who received at least 1 dose of study drug. Only DB period was complete at the time of data cutoff date.
Groups:
- DB Period: Placebo: Participants received crinecerfont-matched placebo orally twice daily for 28 weeks during the DB placebo-controlled treatment period.
- DB Period: Crinecerfont: Participants received crinecerfont orally twice daily for 28 weeks during the DB placebo-controlled treatment period. Dose assignment from Day 1 to Week 28 was based on the participant's weight at Day 1.
Arm/Group | DB Period: Placebo | DB Period: Crinecerfont
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/69
Serious Adverse Events (participants affected / at risk) | 4/33 | 1/69
Other Adverse Events (participants affected / at risk) | 22/33 | 51/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DB Period: Placebo (N=33) | DB Period: Crinecerfont (N=69)
Pyrexia (General disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Chest pain (General disorders) | 1 | 0
Gastroenteritis norovirus (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DB Period: Placebo (N=33) | DB Period: Crinecerfont (N=69)
Headache (Nervous system disorders) | 2 | 17
Pyrexia (General disorders) | 8 | 15
Vomiting (Gastrointestinal disorders) | 8 | 10
Upper respiratory tract infection (Infections and infestations) | 0 | 8
Nasopharyngitis (Infections and infestations) | 6 | 7
Influenza (Infections and infestations) | 2 | 6
Abdominal pain (Gastrointestinal disorders) | 0 | 5
Coronavirus infection (Infections and infestations) | 3 | 5
Fatigue (General disorders) | 0 | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Dizziness (Nervous system disorders) | 3 | 4
Nausea (Gastrointestinal disorders) | 2 | 4
Pharyngitis streptococcal (Infections and infestations) | 0 | 4
Viral infection (Infections and infestations) | 1 | 4
17-hydroxyprogesterone increased (Investigations) | 2 | 3
Blood androstenedione increased (Investigations) | 3 | 3
Blood corticotrophin increased (Investigations) | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 2
Blood insulin increased (Investigations) | 2 | 1
Constipation (Gastrointestinal disorders) | 2 | 1
Tonsillitis (Infections and infestations) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-05-10): https://cdn.clinicaltrials.gov/large-docs/51/NCT04806451/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-18): https://cdn.clinicaltrials.gov/large-docs/51/NCT04806451/SAP_001.pdf